CLINICAL TRIAL: NCT02730507
Title: Surgical Treatment of Spinal Deformity With Sagittal Imbalance Using Patient-specific Rods: A Multicenter, Controlled, Double- Blind Randomized Trial: The PROFILE Study
Acronym: PROFILE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 69HCL14-0444
Record Dates: First submitted 2016-03-23; First posted 2016-04-06 (Estimated); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Spinal Deformity With Sagittal Imbalance
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PSR (Experimental): Bras A : 167 patients in the experimental PSR group. Surgery with patient-specific rod, which are designed according to the preoperative surgical planning of the surgeon in collaboration with the manufacturer.
  Interventions: Device: Surgery with patient-specific rod
- Conventional rod (Active Comparator): Bras B: 167 patients in the experimental conventional rod group
  Interventions: Device: Conventional straight rod

INTERVENTIONS:
Device: Surgery with patient-specific rod — Bras A: PSRs must be used with the appropriate instrumentation designed by the same manufacturer. In order to minimize potential bias derived from using different spinal systems or reduction techniques, the posterior instrumentation must be the same (except the use of standard straight rod) in both groups. The surgical method to implement the PSR will be the same as the one to implement the conventional rod. Except for the bending procedure (patient specific rod or conventional rod with perioperative manual bending), the characteristics of implantable devices (biomaterial and diameter of the rod, design, type of screw, etc.) will be the same in each center.
  Arms: PSR
Device: Conventional straight rod — Bras B: The control group is composed of patients operated with standard straight rods, which are bent in the operating room by the surgeon. In order to minimize potential bias derived from using different spinal systems or reduction techniques, the posterior instrumentation used in the control group must be the same (except the use of PSRs) than the experimental group.
  Arms: Conventional rod

SUMMARY:
Lumbar degenerative diseases (LDD) are an increasingly common condition affecting millions of patients worldwide. LDD can impact not only function, but can also become markedly disabling and cause severe chronic pain. Recent studies support the idea that analysis of sagittal balance is a crucial keypoint to optimize the management of lumbar degenerative diseases, especially when spinal instrumentation is intended.

The first treatment of these pathologies is a medical treatment (medications, physical therapy and exercise). Surgical treatment is frequently necessary if the symptoms worsen and is generally a posterior spinal fusion with instrumentation (screws, hooks and rods) and bone graft. Basic principle of the surgery is to realign the spine along the rod.

Despite documented techniques for surgical planning, it appears that a significant number of patients are ultimately under-corrected after surgery Realignment failure has not only been associated with poor functional outcome but also major complications, such as pseudoarthrosis and rod breakage, which often results in additional surgical procedures.

From a pragmatic point of view, there are two main reasons for realignment failure: poor surgical planning and poor execution. One of the assumptions is that perioperative manual bending of the rod may not always allow the surgeon to restore the sagittal parameters as intended.

A new concept of patient-specific rod (PSR) is now being proposed by a French manufacturer in order to enable an optimal correction and surgical stabilization of the spine. PSR are designed to fit with the patient's unique sagittal spine profile and with surgeons' surgical planning. However, no relevant clinical data is currently available to support the expected medical benefit of this new technology.

The objective of the study is therefore to carry out a study hypothesizing that the use of PSR could improve the percentage of patients whose sagittal profile is optimally corrected after spinal surgery, as well as the patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* • Adult sagittal deformity of the spine defined as

  * a loss of lumbar lordosis versus the pelvic incidence (LL- PI) outside of the range of ±20°
  * PT>25° or SVA>50mm
  * Patients with functional impairment defined as an Oswestry Disability Index over 40/100
  * Spinal posterior fusion and instrumentation indicated for the patient
  * Surgery indicated for 4 or more lumbar levels: from T12 to S1
  * Patients in whom an optimal correction of the sagittal profile is considered to be feasible according to the following criteria:
  * 10°≤ LL-PI≤10°
  * PT < 20°
  * SVA < 40mm.
  * Patients older or equal to 18 years
  * Patients able to sign an informed consent form
  * Patients able to fill out a self-administered questionnaire
  * Patient has to be the beneficiary of the social security system (order n° 2006-477 from April 26th 2006);

Exclusion Criteria:

* • Coronal deformity without sagittal imbalance

  * Patients who required a vertebrectomy
  * Patients who do not required a bone graft or a bone fusion
  * Patient with congenital metabolic bone abnormalities
  * Patient with recent (less than 1month) lumbar vertebrae fracture
  * Patients with insufficient tissue coverage of the surgical site, an insufficient bone quality and quantity.
  * History of an osteoporotic fracture, joint disease with fast evolution, bone resorption, osteopenia
  * Pathologic obesity (BMI > 40)
  * Patients with active or chronic infection, fever or leukocytosis.
  * Suspected or known allergy or intolerance to the medical device used and requesting a combination of different metals.
  * Patient with a medical contraindication to the material used or for which the use of the device could interfere with anatomical structures or expected physiological function.
  * Patients with ongoing treatment of any cancer or history of any cancer of less than 5 years
  * Chronic inflammatory disease
  * Women who are pregnant
  * Patients unable to understand the purpose of the trial or refusing to follow post-surgery instructions.
  * Participation to another trial
  * Patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients whose sagittal profile is optimally corrected between both arms | 12 months.
  The primary end point is the proportion of patients whose sagittal profile is optimally corrected 12 months after a spine-surgery. The optimally corrected sagittal profile definition is based on the following composite criteria:
  * Lombar Lordosis (LL), measured between the superior endplate of L1 and the sacral plate, is equal to the Pelvic Incidence of the patient ± 10° (-10°≤ LL - Pelvic Incidence≤10°)
  * Pelvic Tilt is less than 20°
  * Sagittal Vertical Axis is less than 40mm. These 3 criteria will be measured and combined to define an optimal sagittal profile, by 3 members of an independent committee. Radiographic parameters will be measured on sagittal full-spine x-rays. The patient positioning will be standardized in order to obtain comparable and reproducible images. The positioning is standing both feet on the same alignment, 20-25 cm between the two feet, upper arm fingers tip on the clavicle.

SECONDARY OUTCOMES:
Comparison of the proportion of patients whose sagittal profile is optimally corrected between both arms. | 3 months after surgery
  Same outcome measure as the primary outcome but at different time of follow-up
Comparison of the proportion of patients whose sagittal profile is optimally corrected between both arms. | 6 months after surgery
  Same outcome measure as the primary outcome but at different time of follow-up
Comparison of the proportion of patients whose sagittal profile is optimally corrected between both arms. | 24 months after surgery
  Same outcome measure as the primary outcome but at different time of follow-up

OTHER OUTCOMES:
Comparison of disability index score between both arms. | 3 months after surgery
  Disability index score will be measured using 3 questionnaires: the Owestry disability index, the SRS-22's questionnaire (Scoliosis Research Society) and the Eifel's questionnaire which corresponds to the French version of the Roland and Morris Disability Questionnaire. These three self-questionnaire will be proposed to each participant at the 3, 6, 12 and 24 months visit of follow-up
Comparison of disability index score between both arms. | 6 months after surgery
  Disability index score will be measured using 3 questionnaires: the Owestry disability index, the SRS-22's questionnaire (Scoliosis Research Society) and the Eifel's questionnaire which corresponds to the French version of the Roland and Morris Disability Questionnaire. These three self-questionnaire will be proposed to each participant at the 3, 6, 12 and 24 months visit of follow-up
Comparison of disability index score between both arms. | 12 months after surgery
  Disability index score will be measured using 3 questionnaires: the Owestry disability index, the SRS-22's questionnaire (Scoliosis Research Society) and the Eifel's questionnaire which corresponds to the French version of the Roland and Morris Disability Questionnaire. These three self-questionnaire will be proposed to each participant at the 3, 6, 12 and 24 months visit of follow-up
Comparison of disability index score between both arms. | 24 months after surgery
  Disability index score will be measured using 3 questionnaires: the Owestry disability index, the SRS-22's questionnaire (Scoliosis Research Society) and the Eifel's questionnaire which corresponds to the French version of the Roland and Morris Disability Questionnaire. These three self-questionnaire will be proposed to each participant at the 3, 6, 12 and 24 months visit of follow-up
Comparison of pain level between both arms. | 6 months after surgery
  Pain relief will be measured using a Visual Analogic Scale at 6, 12, 24 months
Comparison of pain level between both arms. | 12 months after surgery
  Pain relief will be measured using a Visual Analogic Scale at 6, 12, 24 months
Comparison of pain level between both arms. | 24 months after surgery
  Pain relief will be measured using a Visual Analogic Scale at 6, 12, 24 months
Comparison of radiographic sagittal parameters measured on sagittal full-spine x-rays | 3 months after surgery
  Several radiographic parameters such as Pelvic incidence, Lumbar lordosis, Real lordosis, Thoracic kyphosis, Real thoracic kyphosis, Sagittal vertical axis, Pelvic tilt, Spino-sacral angle and C7 plumb line /Sacro-femoral distance. The patients will be in a standing position when taking an x-ray. The Full spine X-Ray should include at least from C7 to femoral heads (proximal part of the femur) from both AP and lateral profiles.
Comparison of radiographic sagittal parameters measured on sagittal full-spine x-rays | 6 months after surgery
  Several radiographic parameters such as Pelvic incidence, Lumbar lordosis, Real lordosis, Thoracic kyphosis, Real thoracic kyphosis, Sagittal vertical axis, Pelvic tilt, Spino-sacral angle and C7 plumb line /Sacro-femoral distance. The patients will be in a standing position when taking an x-ray. The Full spine X-Ray should include at least from C7 to femoral heads (proximal part of the femur) from both AP and lateral profiles.
Comparison of radiographic sagittal parameters measured on sagittal full-spine x-rays | 12 months after surgery
  Several radiographic parameters such as Pelvic incidence, Lumbar lordosis, Real lordosis, Thoracic kyphosis, Real thoracic kyphosis, Sagittal vertical axis, Pelvic tilt, Spino-sacral angle and C7 plumb line /Sacro-femoral distance. The patients will be in a standing position when taking an x-ray. The Full spine X-Ray should include at least from C7 to femoral heads (proximal part of the femur) from both AP and lateral profiles.
Comparison of radiographic sagittal parameters measured on sagittal full-spine x-rays | 24 months after surgery
  Several radiographic parameters such as Pelvic incidence, Lumbar lordosis, Real lordosis, Thoracic kyphosis, Real thoracic kyphosis, Sagittal vertical axis, Pelvic tilt, Spino-sacral angle and C7 plumb line /Sacro-femoral distance. The patients will be in a standing position when taking an x-ray. The Full spine X-Ray should include at least from C7 to femoral heads (proximal part of the femur) from both AP and lateral profiles.
Comparison of the proportion of peri- and postoperative complications | intraoperative and the follow-up visit at 3 month
  Frequency of peri- and postoperative adverse events related to the device (especially a rod breakage) or the surgery
Comparison of the proportion of peri- and postoperative complications | intraoperative and the follow-up visit at 6 month
  Frequency of peri- and postoperative adverse events related to the device (especially a rod breakage) or the surgery
Comparison of the proportion of peri- and postoperative complications | intraoperative and the follow-up visit at 12 month
  Frequency of peri- and postoperative adverse events related to the device (especially a rod breakage) or the surgery
Comparison of the proportion of peri- and postoperative complications | intraoperative and the follow-up visit at 24 month
  Frequency of peri- and postoperative adverse events related to the device (especially a rod breakage) or the surgery
Time of procedure evaluation | intraoperative
  Comparison of the duration in minutes of the rod bending time in the operating room

CONTACTS AND LOCATIONS:
Overall Officials: Cedric BARREY, PHD, Study Director — Hospices Civils de Lyon

IPD SHARING:
Plan to Share IPD: No